CLINICAL TRIAL: NCT03260946
Title: The Use of Complementary Medicine in Palliative/Supportive Care Centres in Lyon, France
Brief Title: The Use of Alternative Medicine by Palliative Care Patients
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0217
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2017-08

CONDITIONS: Cancer; Terminal Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palliative/Supportive care: Individuals with cancer receiving palliative or supportive care
  Interventions: Other: Complementary medicine use

INTERVENTIONS:
Other: Complementary medicine use — The prevalence of complementary medicine use

SUMMARY:
Palliative care centres in Lyon, France as well as the disclosure of Complementary and Alternative Medicine and conventional healthcare use to conventional and Complementary and Alternative Medicine practitioners respectively.

These aims will be achieved through the following objectives:

1. Describe the prevalence of Complementary and Alternative Medicine practitioner and product use in the outpatient population of palliative care centres in Lyon, France
2. Describe the characteristics of Complementary and Alternative Medicine users the outpatient population of palliative care centres in Lyon, France
3. Estimate the Complementary and Alternative Medicine expenditure of the outpatient population of palliative care centres in Lyon, France
4. Describe the rates of disclosure of both Complementary and Alternative Medicine and conventional health care to health professionals by the outpatient population of palliative care centres in Lyon, France
5. Describe the reasons for disclosure or non-disclosure of both Complementary and Alternative Medicine and conventional health care to health professionals by the outpatient population of palliative care centres in Lyon, France

ELIGIBILITY:
Inclusion Criteria:

1. Patients accessing care from a palliative/supportive care centre in Lyon, France
2. Can read and understand French
3. Has been diagnosed with cancer

Exclusion Criteria:

1. The primary health condition for which they are attending the centre is not cancer
2. They are not able to read and understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with cancer receiving palliative or supportive care
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Complementary medicine use | 15 minutes
  The prevalence of complementary medicine use. Data collected using a questionnaire.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - USP de Charmettes - Croix rouge française, Lyon
  - Service E.M.S.P. Groupement Hospitalier Nord - Hôpital de la Croix-Rousse, Lyon
  - Centre de Soins Palliatifs Lyon-Sud Pavillon 1K - Centre Hospitalier Lyon-Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No